CLINICAL TRIAL: NCT03662958
Title: Evaluation of the Testosterone Suppressive Effect in Healthy Male Volunteers of a Novel Leuprolide Acetate 3.75mg Depot (Lutrate) VS Market Reference Leuprolide Acetate 3.75mg Depot (Enantone)
Brief Title: Comparison of a Novel Leuprolide With Market Leuprolide
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Lee's Pharmaceutical Limited (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: ZK-LUT-201802
Record Dates: First submitted 2018-08-30; First posted 2018-09-10 (Actual); Last update posted 2018-09-10 (Actual); Status verified 2018-09

CONDITIONS: Prostate Cancer
MeSH Terms: conditions — Prostatic Neoplasms | interventions — Leuprolide

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Lutrate (Experimental): a novel leuprolide acetate 3.75mg depot
  Interventions: Drug: Lutrate
- Enantone (Active Comparator): market reference leuprolide acetate 3.75 mg depot
  Interventions: Drug: Enantone

INTERVENTIONS:
Drug: Lutrate — a novel leuprolide acetate 3.75mg depot
  Arms: Lutrate
Drug: Enantone — market reference leuprolide acetate 3.75 mg depot
  Arms: Enantone

SUMMARY:
This is a single dose, randomized, single blind, parallel group study to evaluate the testosterone suppressive effect in healthy male volunteers of a novel leuprolide acetate 3.75mg depot vs market reference leuprolide acetate 3.75mg depot. The safety, tolerability and the pharmacokinetic properties of the investigational drug and the control drug will also be assessed.

ELIGIBILITY:
Inclusion Criteria:

1. Males of 18-40 years old (inclusive). The age difference of subjects within and between groups should be less than 10 years, at the time of screening.
2. Body weight of at least 50kg. BMI to be 19-24 kg/m2 (inclusive).
3. Able to comprehend the full nature and purpose of the study, including potential risks and side effects; able to cooperate with investigators and to comply with the requirements of the study
4. Signed informed consent form prior to any screening procedures

Exclusion Criteria:

1. Clinically significant and relevant history of cardiovascular, hepatic, renal, hematologic, endocrine, respiratory, neurological diseases or acute/chronic diseases of the digestive tract.
2. History of hypersensitivity towards leuprolide, synthetic LHRH or LHRH derivatives or any excipients of the study formulation.
3. Abnormal and clinically significant 12-lead ECG
4. Abnormal and clinically significant laboratory assessments
5. Blood donation or blood loss greater than or equal to 400mL within 3 months prior to screening
6. Participation of clinical trials within 3 months prior to screening
7. Use of any drugs within 2 weeks prior to screening
8. History of drug abuse within 1 year prior to screening
9. History of alcohol abuse within 1 years prior to screening
10. History of tobacco smoking (more than 5 cigarette per day) within 1 year prior to screening
11. Abnormal testosterone level at screening (not in the range of 168-781ng/dL)
12. Dermatitis or skin anomalies that might affect the administration area and the surroundings
13. Subject or his partner not willing to adopt appropriate contraceptive measures
14. Subjects have a history of depressive illness or sexual dysfunction;
15. Subjects that the investigator deems unsuitable to be enrolled
16. Subject not willing to cooperate with the investigators.

Ages: 18 Years to 40 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 48 (Estimated)
Dates: Start 2018-08-01 (Actual); Primary Completion 2018-10 (Estimated); Study Completion 2018-12 (Estimated)

PRIMARY OUTCOMES:
The rate of castration at the end of week 4 (i.e. day 29) | 4 weeks

SECONDARY OUTCOMES:
The time to castration (i.e Tlag) between the 2 groups after administration of leuprolide | 4 weeks
The duration of castration (i.e Tcast) | 4 weeks
LH concentration | 4 weeks
FSH concentration | 4 weeks

OTHER OUTCOMES:
Adverse events | 4 weeks
Local tolerability | post-dose 5 min and 1 hour, day 8, 15 and 29
  (10) Subjects will evaluate pain with VAS. Investigators will evaluate redness and induration with a 4-point scale.
AE | 4 weeks
blood pressure | 4 weeks
pulse rate | 4 weeks
respiratory rate | 4 weeks
body temperature | 4 weeks
12-lead ECG | 4 weeks
body weight | 4 weeks

CONTACTS AND LOCATIONS:
Locations (1):
- The First Affiliated Hospital of Bengbu Medical College, Bengbu, Anhui, China

IPD SHARING:
Plan to Share IPD: Undecided